CLINICAL TRIAL: NCT05245799
Title: "Effectiveness of Adding a Novel Digital Storybook Intervention Platform in Therapy to Improve Speech, Language, and Literacy Outcomes in Children With Hearing Loss"
Brief Title: Hear Me Read 2021 Clinical Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Prasanth Pattisapu (Other)
Collaborators: Clinical and Translational Intramural Funding Program from the Abigail Wexner Research Institute (Unknown)
Responsible Party: Sponsor-Investigator, Prasanth Pattisapu, Principal Investigator, Nationwide Children's Hospital
Organization: Nationwide Children's Hospital (Other)
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00001863; AWD00001881 (Other Grant/Funding Number: IFPAWRI)
Record Dates: First submitted 2022-01-14; First posted 2022-02-18 (Actual); Last update posted 2023-03-30 (Actual); Status verified 2023-03

CONDITIONS: Hearing Loss; Deafness; Hearing Disorders in Children; Hearing Impaired Children; Speech Therapy; Speech Disorders in Children; Literacy
Keywords: App; Speech and Language; Tablet; Digital; Literacy; Hearing Loss; Speech Therapy
MeSH Terms: conditions — Hearing Loss; Deafness; Communication Disorders; Literacy; Alzheimer Disease; Speech; Language | interventions — Speech Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Speech Language Therapy (Active Comparator): Children who are deaf/hard of hearing will receive standard of care speech and language therapy with a speech language pathologist. Reading time is prescribed 20 min, 3x/week.
  Interventions: Behavioral: Speech Language Therapy
- Speech Language Therapy + Digital Phase (Experimental): Children who are deaf/hard of hearing will receive standard of care speech and language therapy with a speech language pathologist with the addition of the digital app named, Hear Me Read, that will be used to achieve reading, speech and language goals through interactive digital storybook reading. Reading time is prescribed 20 min, 3x/week.
  Interventions: Behavioral: Speech Language Therapy; Behavioral: Digital Software Application

INTERVENTIONS:
Behavioral: Speech Language Therapy — Children who are deaf/hard of hearing will receive typical speech and language therapy with a speech pathologist. Reading time is prescribed 20 min, 3x/week.
Behavioral: Digital Software Application — The Hear Me Read app is an IOS-based software application that enables parents and speech-language pathologists to partner together to help deaf/hard of hearing children (D/HH) achieve reading, speech and language goals through interactive digital storybook reading.
  Other Names: Hear Me Read
  Arms: Speech Language Therapy + Digital Phase

SUMMARY:
The purpose of this study is to evaluate if the effects of in-person speech-language therapy with a novel digital storybook intervention platform (Hear Me Read) improves vocabulary, speech and language, and literacy outcomes in young children who are deaf or hard of hearing compared with in-person therapy alone.

DETAILED DESCRIPTION:
For this study, 50 children, who are deaf/hard of hearing, and their caregiver will be enrolled into 2 separate 6-month intervention periods, for a total of 12 months of participation. There are two intervention periods in this study, Intervention Period 1 (SLT) and Intervention Period 2 (SLT+Digital). Each one lasts about 6 months and every participant will participate in both intervention periods.

Intervention Period 1 is the speech-language therapy (SLT) only intervention. During this intervention, the child will go to speech therapy as normally prescribed by their speech language pathologist. There will be standardized reading time that is prescribed at 20 minutes, 3 times a week and will be completed at home by the child and caregiver.

Intervention Period 2 is the speech-language therapy with the Hear Me Read (SLT+Digital) intervention. During this intervention, the child will continue to go to speech therapy as they typically would, but will be asked to use the Hear Me Read app. There will be standardized reading time that is prescribed at 20 minutes, 3 times a week and will be completed at home by the child and caregiver using the Hear Me Read app.

ELIGIBILITY:
Inclusion Criteria:

* Male and female children ages 3.0-5.11 (5 years and 11 months) at time of initial assessment and:
* Bilateral Sensorineural or mixed hearing loss at least (PTA≥30dB)
* Auditory neuropathy in both ears

Exclusion Criteria:

* English not primary language
* Standard score CLS >2 SD from normal on CELF-P3

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2022-03-25 (Actual); Primary Completion 2024-03-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Receptive One Word Picture Vocabulary Test | 12- month intervention period
  The ROWPVT-4 is an individually administered assessment of how well persons can match a word that is heard to objects, actions, or concepts presented in full-color pictures. The examinee indicates the correct color picture that matches the word spoken by the examiner. Raw scores are reported as standard scores, percentile ranks, growth scale and age equivalents. Raw scores are from 0-100 with higher scores indicating better performance.
Clinical Evaluation of Language Fundamentals Preschool- 3 and subtests: Sentence Comprehension | 12- month intervention period
  The Sentence Comprehension (SC) subtest is used to evaluate the child's ability to interpret spoken sentences of increasing length and complexity. The child identifies a picture that matches the sentence read aloud by the examiner. Raw scores (min = 0; max = 22) are reported as standard scores, percentile ranks, growth scale and age equivalents. Higher scaled scores represent better language outcomes.
Clinical Evaluation of Language Fundamentals Preschool- 3 and subtests: Word Structure | 12- month intervention period
  The Word Structure (WS) subtest is used to evaluate the child's ability to (a) apply word structure rules to mark inflections, derivations, and comparison and (b) select and use appropriate pronouns to refer to people, objects, and possessive relationships. Raw scores (min = 0; max = 24) are reported as standard scores, percentile ranks, growth scale and age equivalents. Higher standard scores represent better language outcomes.
Clinical Evaluation of Language Fundamentals Preschool- 3 and subtests: Expressive Vocabulary | 12- month intervention period
  The Expressive Vocabulary (EV) subtest is used to evaluate the child's ability to label images of people, objects, attributes, and actions. The child names an object, person, or activity portrayed in a picture. Raw scores (min = 0; max = 42) are reported as standard scores, percentile ranks, growth scale and age equivalents. Higher standard scores represent better language outcomes.
Clinical Evaluation of Language Fundamentals Preschool- 3 and subtests: Following Directions | 12- month intervention period
  The Following Directions (FD) subtest is used to evaluate the child's ability to (a) interpret spoken directions of increasing length and complexity; (b) remember the names, characteristics, and order of mention of pictures; and (c) identify the targets from among several choices. Raw scores (min = 0; max = 24) are reported as standard scores, percentile ranks, growth scale and age equivalents. Higher standard scores represent better language outcomes.
Clinical Evaluation of Language Fundamentals Preschool- 3 and subtests: Recalling Sentences | 12- month intervention period
  The Recalling Sentences (RS) subtest is used to evaluate the child's ability to listen to spoken sentences of increasing length and complexity and repeat the sentences without changing word meanings, inflections, derivations or comparisons, or sentence structure. Raw scores (min = 0; max = 45) are reported as standard scores, percentile ranks, growth scale and age equivalents. Higher standard scores represent better language outcomes.
Clinical Evaluation of Language Fundamentals Preschool- 3 and subtests: Basic Concepts | 12- month intervention period
  The Basic Concepts (BC) subtest is used to evaluate the child's knowledge of concepts including direction/location/position, number/quantity, sequence, attributes, dimension/size, same/different, and inclusion/exclusion. Raw scores (min = 0; max = 24) are reported as standard scores, percentile ranks, growth scale and age equivalents. Higher standard scores represent better language outcomes.
Clinical Evaluation of Language Fundamentals Preschool- 3 and subtests: Word Classes | 12- month intervention period
  The Word Classes (WC) subtest is used to evaluate the child's ability to perceive relationships between words that are related by semantic class features. Raw scores (min = 0; max = 20) are reported as standard scores, percentile ranks, growth scale and age equivalents. Higher standard scores represent better language outcomes.
Clinical Evaluation of Language Fundamentals Preschool- 3: Core Language Score | 12- month intervention period
  The Core Language Score (CLS) is a measure of general language ability that quantifies overall language performance and is used to make decisions about the presence or absence of a language disorder. It is derived by summing the scaled scores from the subtests that best discriminate typical language performance from disordered language performance deriving a standardized composite score (min = 45; max = 155). Higher composite scores represent better language outcomes.
Clinical Evaluation of Language Fundamentals Preschool- 3 and Indices: Receptive Language Index | 12- month intervention period
  The Receptive Language Index (RLI) is a measure of listening and auditory comprehension and is derived by summing the scaled scores from a combination of two or three receptive subtests. Scores are derived by summing the scaled scores from the subtests and deriving a standardized composite score (min = 45; max = 155). Higher composite scores represent better language outcomes.
Clinical Evaluation of Language Fundamentals Preschool- 3 and Indices: Expressive Language Index | 12- month intervention period
  The Expressive Language Index (ELI) is a measure of performance on three tests that probe expressive aspects of language including oral language expression. Scores are derived by summing the scaled scores from the subtests and deriving a standardized composite score (min = 45; max = 155). Higher composite scores represent better language outcomes.

SECONDARY OUTCOMES:
Clinical Evaluation of Language Fundamentals Preschool- 3 and subtests: Phonological Awareness | 12- month intervention period
  The Phonological Awareness (PA) subtest is used to evaluate the child's knowledge of the sound structure of language and ability to manipulate sound through compound word and syllable blending, sentence and syllable segmentation, and rhyme awareness and production. Raw scores (min = 0; max = 24) are reported as standard scores, percentile ranks, growth scale and age equivalents. Higher standard scores represent better language outcomes.
Clinical Evaluation of Language Fundamentals Preschool- 3 and subtests: Preliteracy Rating Scale | 12- month intervention period
  The Preliteracy Rating Scale (PRS) subtest is used to identify preliteracy skills that may influence development of reading and writing skills. The examiner provides or elicits information from a respondent about the child's early reading and writing skills. Raw scores (min = 0; max = 105) are reported as standard scores, percentile ranks, growth scale and age equivalents. Higher standard scores represent better language outcomes.
Clinical Evaluation of Language Fundamentals Preschool-3 Index: Early Literacy Index | 12- month intervention period
  Early Literacy Index (ELI) is a measure of performance on two subtests designed to assess early literacy skills. Scores are derived by summing the scaled scores from the subtests and deriving a standardized composite score (min = 45; max = 155). Higher composite scores represent better language outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Prasanth Pattisapu, MD, Principal Investigator — Nationwide Children's Hospital
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No